CLINICAL TRIAL: NCT04323683
Title: The Effect of Progesterone Levels on Human Endometrial Transcriptomics During the Implantation Window
Brief Title: The Effect of Progesterone on Human Endometrium
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Walid Maalouf, Course Director MMedSci Assisted Reproduction Technology, Faculty of Medicine & Health Sciences, University of Nottingham
Other Study IDs: 13/EM/0277
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Fertility
MeSH Terms: interventions — Gene Expression Profiling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA obtained from endometrium
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low progesterone: Women with progesterone level below 15 ng/ml
  Interventions: Genetic: Microarray
- Normal progesterone: Women with progesterone level above 15 ng/ml
  Interventions: Genetic: Microarray

INTERVENTIONS:
Genetic: Microarray — High throughput technique for determining global gene expression of the condition of interest

SUMMARY:
This study evaluates the relationship between progesterone levels and endometrial gene expression

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-35, regular menstrual cycles, the cycle length between 25 and 35 days, body mass index (BMI) between 18 - 25

Exclusion Criteria:

* History of infertility, history of pelvic pain or/and endometriosis, history of pelvic mass, history of hormonal therapy in the last 3 months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fertile women
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Differentially expressed genes between women with low and normal progesterone | 2 months
  Fold-change and p-value were used to determine differentially expressed genes using Partek software

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's medical center, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No